CLINICAL TRIAL: NCT04479904
Title: A Single-Arm, Open-Label, Multi-Center, Phase II Study of Famitinib Malate to Treat Intrahepatic Cholangiocarcinoma Patients With FGFR2(Fibroblast Growth Factor Receptor2) Genetic Aberrations Who Failed First-Line Therapy
Brief Title: A Trial of Famitinib in Patients With Failure of First-Line Treatment For Intrahepatic Cholangiocarcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: It is difficult to screening subject
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1020-II-204
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2020-07

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — famitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- famitinib (Experimental)
  Interventions: Drug: Famitinib

INTERVENTIONS:
Drug: Famitinib — po

SUMMARY:
This is a single-arm, open-label, multi-center Phase II clinical trial intended to observe and evaluate the efficacy and safety of famitinib malate in treating iCCA(Intrahepatic Cholangiocarcinoma ) patients with FGFR2 genetic aberrations who failed first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent;
2. Aged 18-75 years (inclusive), males and females;
3. Those with histopathologically diagnosed iCCA, who had previously undergone but failed first-line systematic chemotherapy;
4. FGFR2 fusion/rearrangement confirmed by tests conducted in designated central laboratory;
5. At least one measurable lesion that has not been treated locally;
6. ECOG score of 0-1;
7. Expected survival ≥ 12 weeks;

Exclusion Criteria:

1. Presence of multiple factors affecting oral medications;
2. Wounds unhealed over a long period of time, or fractures not completely healed;
3. Known or suspected allergy to investigational drug or any drug related to this trial.
4. Known cases of CNS(Central Nervous System) metastasis;
5. Uncontrolled cardiac diseases or symptoms;
6. Patients with congenital or acquired immunodeficiency (such as HIV positive), or a history of organ transplants;
7. Patients previously treated with FGFR inhibitors (such as erdafitinib)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-10 (Estimated); Primary Completion 2021-12-10 (Estimated); Study Completion 2022-02-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate per RECIST 1.1 | up to 24 months

SECONDARY OUTCOMES:
DOR | At pre-defined intervals from initial dose up to 24 months
  Duration of Response
DCR | At pre-defined intervals from initial dose up to 24 months
  Disease Control Rate
PFS | At pre-defined intervals from initial dose up to 24 months
  Progression-Free-Survival
OS | At pre-defined intervals from initial dose up to 24 months
  Overall survival
Adverse events (AE) and serious adverse event (SAE) | At pre-defined intervals from initial dose up to 24 months
  Including incidence, grade (according to CTCAE V5.0 criteria), severity, duration, and causality with investigational drug
Plasma concentrations of famitinib and its N-desethyl metabolite | At pre-defined intervals from initial dose up to 24 months